CLINICAL TRIAL: NCT04010253
Title: Impact of Bronchial Drainage by the Medical Device Simeox® on Function and Respiratory Symptoms Compared to Manual Autogenous Drainage Physiotherapy in Adult Cystic Fibrosis Patients
Brief Title: Impact of Bronchial Drainage Technique by the Medical Device Simeox® on Respiratory Function and Symptoms in Adult Patients With Cystic Fibrosis
Acronym: MUCOSIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A00622-55
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Physiotherapy; Drainage
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIMEOX (Experimental)
  Interventions: Other: Autogenic drainage
- Autogenic Drainage (Active Comparator)
  Interventions: Device: SIMEOX

INTERVENTIONS:
Device: SIMEOX — Instrumental airway clearance by the medical device SIMEOX
  Arms: Autogenic Drainage
Other: Autogenic drainage — Manual aiway clearance by autogenic drainage
  Arms: SIMEOX

SUMMARY:
The main objective of the study is to evaluate the short-term effects of the airway clearance technique by the medical device Simeox (Physio Assist, France) versus Autogenic Drainage, on the pulmonary function of adult patients with stable cystic fibrosis. To analyse these effects, the investigators used forced oscillation technique measured by TremoFlo™ C-100 Airwave Oscillometry System™ (THORASYS Thoracic Medical Systems Inc. Montreal, Quebec, Canada) with an evaluation of the perceived clinical benefits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis confirmed
* Age ≥18 years
* 30% <FEV1 <70% predicted
* Presence of bronchial congestion reported by the patient or the investigator

Exclusion Criteria:

* Uncontrolled asthma
* Pneumothorax <6 weeks
* Recent severe hemoptysis <6 weeks
* Patient registered on the transplant list
* Exacerbation within 4 weeks (3 months if hospitalization) before screening
* Cardiovascular disorders, electrocardiogram (ECG) parameters or clinically significant respiratory (non-cystic fibrosis) conditions
* Patients unable to perform measurements of ROF, spirometry, plethysmography.
* Any contraindication to manual or instrumental physiotherapy.
* Pregnancy, breastfeeding.
* Patient under tutorship or curatorship
* No affiliation to the French social security
* Patient using Simeox at home
* Patient under Trikafta for less than 6 weeks.
* Patient using Simeox more than twice a week during physiotherapy sessions, not wanting a washout period of 7 days before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Low frequency resistance R5 | 1 month
  Comparison of variations V4 and V8 sessions (pre and post airway clearance session)

SECONDARY OUTCOMES:
Comparison of the impact of Simeox® bronchial drainage compared to autogenous drainage on respiratory symptoms: dyspnea, congestion and fatigue | 1 month
Evaluation of the distal and / or proximal decluttering by the two techniques, according to the improvement profile of the forced oscillations | 1 month
Evaluation of the impact of Simeox® bronchial drainage vs autogenous drainage by spirometry and plethysmography (distension and resistance) | 1 month
Evaluation of correlations between clinical benefit and changes in functional respiratory investigations (forced oscillations, spirometry, plethysmography) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PEREZ, MD, Principal Investigator — CHRU LILLE
Locations (8):
- France (8):
  - CH Amiens, Amiens
  - Hôpital la Bocage CHRU de Dijon, Dijon
  - CHRU Lille - Hopital Calmette, Lille
  - GH Sud - Hospices Civils de Lyon, Lyon
  - CH Nice, Nice
  - Soins de Suite Nutritionnels et Respiratoires -Fondation IDLYS, Roscoff
  - CHU de Rouen, Rouen
  - Hopital Larrey, Toulouse